CLINICAL TRIAL: NCT04225273
Title: Open Label Extension Study for 43USSA1705 (A Randomized, Evaluator-blinded, Multi-center Study to Evaluate the Safety and Effectiveness of Sculptra Aesthetic for Correction of Nasolabial Folds)
Brief Title: Extension Study for 43USSA1705
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43USSA1705ext
Record Dates: First submitted 2019-12-04; First posted 2020-01-13 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Sculptra Aesthetic (Experimental): Participants who completed 48 weeks of Sculptra Aesthetic reconstituted with 8 milliliters (mL) of sterile water for injection (SWFI) in study 43USSA1705 (NCT03780244) were followed into this long-term extension study at Week 72 and Week 96 after baseline (i.e., Day 1/first treatment session with Sculptra Aesthetic in Study 43USSA1705 [NCT03780244]). No investigational product was provided during this extension study.
  Interventions: Device: Sculptra Aesthetic, Lidocaine HCL

INTERVENTIONS:
Device: Sculptra Aesthetic, Lidocaine HCL — No intervention was administered during this extension study.

SUMMARY:
To evaluate the long-term safety of Sculptra Aesthetic as a single regimen for correction of Nasolabial Fold (NLF) contour deficiencies after changes in reconstitution and injection procedures compared to the approved label.

ELIGIBILITY:
Inclusion Criteria:

* Randomized to Sculptra Aesthetic 8ml reconstitution and successfully completed study 43USSA1705

Exclusion Criteria:

* Medical condition that in the opinion of the Investigator would make the subject unsuitable for inclusion
* Other condition preventing the subject from entering the study in the Investigator's opinion
* Participation in any interventional clinical study throughout the duration of the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Galderma Study Site, Scottsdale, Arizona
  - Galderma Study Site, Bradenton, Florida
  - Galderma Study Site, Austin, Texas
  - Galderma Study Site, Spring, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 38 participants entered this long-term extension study upon completion of Study 43USSA1705 (NCT03780244) (Week 48) and performed follow-up visits in this extension study at Week 72 and Week 96 after baseline (that is [i.e.], Day1/first treatment session in Study 43USSA1705 [NCT03780244]). No treatment was given during this extension study.
Period: Overall Study
Arm/Group | Sculptra Aesthetic
Started | 38
Completed | 35
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: The extension population included all participants who entered the extension study. Baseline was defined as the observation that was closest to but prior to study treatment at the baseline visit/first treatment in Study 43USSA1705 (NCT03780244).
Groups:
- Sculptra Aesthetic: Participants who completed 48 weeks of Sculptra Aesthetic reconstituted with 8 mL of SWFI in study 43USSA1705 (NCT03780244) were followed into this long-term extension study at Week 72 and Week 96 after baseline (i.e., Day 1/first treatment session with Sculptra Aesthetic in Study 43USSA1705 [NCT03780244]). No investigational product was provided during this extension study.
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38
Fitzpatrick Skin Type (FST) [Count of Participants; unit: Participants] — FST is a numerical classification scale for the color of skin from Type I to Type VI. Type I= always burns, never tans; Type II= usually burns, tans minimally (light colored but darker than fair); Type III= sometimes mild burn, tans uniformly (golden honey or olive); Type IV= burns minimally, always tan well (moderate brown); Type V= very rarely burns, tans very easily (dark brown); Type VI= never burns (deeply pigmented dark brown to darkest brown). A higher type was considered better.
  Participants
    FST I | 2
    FST II | 7
    FST III | 16
    FST IV | 6
    FST V | 5
    FST VI | 2
Baseline Wrinkle Assessment Scale (WAS) (Left) [Mean (Standard Deviation); unit: units on a scale] — The WAS is a validated photograph-based outcome instrument that is designed specifically for quantifying facial folds. Scoring of nasolabial fold (NLF) wrinkle severity (grades 0-5, with 0 representing no wrinkles and 5 representing very deep wrinkles, redundant fold) was based on visual live assessment by the Blinded Evaluator. Lower scores indicate better outcome.
  units on a scale | 3.0 (0.70)
Baseline WAS (Right) [Mean (Standard Deviation); unit: units on a scale] — The WAS is a validated photograph-based outcome instrument that is designed specifically for quantifying facial folds. Scoring of NLF wrinkle severity (grades 0-5, with 0 representing no wrinkles and 5 representing very deep wrinkles, redundant fold) was based on visual live assessment by the Blinded Evaluator. Lower scores indicate better outcome.
  units on a scale | 2.8 (0.79)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Both Sides of the Face as Assessed by the Evaluator Using the WAS at Weeks 72 and 96
Description: The WAS is a validated photograph-based outcome instrument that is designed specifically for quantifying facial folds. Scoring of NLF wrinkle severity (grades 0-5, with 0 representing no wrinkles and 5 representing very deep wrinkles, redundant fold) was based on visual live assessment by the Blinded Evaluator at defined timepoints. Lower scores indicate better outcome. Effectiveness is defined as change from baseline on both sides of the face using WAS at 72 and 96 weeks after the first treatment session. Baseline was defined as the observation that was closest to but prior to study treatment at the baseline visit/first treatment in Study 43USSA1705 (NCT03780244). Therefore, Weeks 72 and 96 in timeframe represents timepoints of current extension study and calculated from baseline of 43USSA1705 (NCT03780244).
Time Frame: Baseline of study 43USSA1705 (NCT03780244), Weeks 72 and 96 (assessed in the current extension study)
Population: The extension population included all participants who entered the extension study. Here, "overall number of participants analyzed" refers to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome measure at given timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
units on a scale
  Left NLF: Change at Week 72: number analyzed (Participants) | 34
  Left NLF: Change at Week 72 | -1.3 (1.06)
  Right NLF: Change at Week 72: number analyzed (Participants) | 34
  Right NLF: Change at Week 72 | -1.2 (0.88)
  Left NLF: Change at Week 96 | -1.2 (1.13)
  Right NLF: Change at Week 96 | -1.1 (1.08)

2. Secondary Outcome: Number of Participants (Responders) Assessed Using the Global Aesthetic Improvement Scale (GAIS) Based on the Participants Live Assessment
Description: A responder was defined as a participant assessed as at least "Improved" (very much improved, much improved, and improved) on both sides of the face concurrently assessed using GAIS by participant. The 7-graded GAIS used by the participant to live assess the aesthetic improvement had responses as follows: (3) Very Much Improved, (2) Much Improved, (1) Improved, (0) No Change, (-1) Worse, (-2) Much Worse, and (-3) Very Much Worse. For reporting of outcomes, the higher the GAIS value, the greater the improvement (Range -3 to 3). Baseline was defined as the observation that was closest to but prior to study treatment at the baseline visit/first treatment in Study 43USSA1705 (NCT03780244). Therefore, Weeks 72 and 96 in timeframe represents timepoints of current extension study and calculated from baseline of 43USSA1705 (NCT03780244).
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: The extension population included all participants who entered the extension study. Here, "overall number of participants analyzed" refers to the participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72 | 30
  Week 96 | 30

3. Secondary Outcome: Number of Participants (Responders) Assessed Using the GAIS Based on the Investigator Live Assessment
Description: A responder was defined as a participant assessed as at least "Improved" (very much improved, much improved, and improved) on both sides of the face concurrently assessed using GAIS by investigator. The 7-graded GAIS used by the participant to live assess the aesthetic improvement had responses as follows: (3) Very Much Improved, (2) Much Improved, (1) Improved, (0) No Change, (-1) Worse, (-2) Much Worse, and (-3) Very Much Worse. For reporting of outcomes, the higher the GAIS value, the greater the improvement (Range -3 to 3). Baseline was defined as the observation that was closest to but prior to study treatment at the baseline visit/first treatment in Study 43USSA1705. (NCT03780244). Therefore, Weeks 72 and 96 in timeframe represents timepoints of current extension study and calculated from baseline of 43USSA1705 (NCT03780244).
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72 | 35
  Week 96 | 35

4. Secondary Outcome: FACE-Q™ Appraisal of Lines Rasch Transformed Total Scores: NLF Questionnaire
Description: FACE-Q™ appraisal of lines NLF scores were used to assess participant's treatment satisfaction. The sum of the participants FACE-Q™ appraisal of lines NLF scores was converted to a Rasch-transformed total score (ranged from 0 to 100) according to the FACE-Q™ manual; a higher total score indicated greater participant satisfaction. Baseline was defined as the observation that was closest to but prior to study treatment at the baseline visit/first treatment in Study 43USSA1705. (NCT03780244). Therefore, Weeks 72 and 96 in timeframe represents timepoints of current extension study and calculated from baseline of 43USSA1705 (NCT03780244).
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
score on a scale
  Week 72 | 69.8 (25.05)
  Week 96 | 70.2 (25.46)

5. Secondary Outcome: Subject Satisfaction With Treatment: Would You Recommend the Treatment to a Friend?
Description: A subject satisfaction question with responses Yes or No. Baseline was defined as the observation that was closest to but prior to study treatment at the baseline visit/first treatment in Study 43USSA1705 (NCT03780244). Therefore, Weeks 72 and 96 in timeframe represents timepoints of current extension study and calculated from baseline of 43USSA1705 (NCT03780244).
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Yes | 33
  Week 72: No | 2
  Week 96: Yes | 31
  Week 96: No | 4

6. Secondary Outcome: Subject Satisfaction With Treatment: Would You do the Treatment Again?
Description: as for outcome 5
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Yes | 32
  Week 72: No | 3
  Week 96: Yes | 32
  Week 96: No | 3

7. Secondary Outcome: Subject Satisfaction With Treatment: Would You Say the Subtle Treatment Results Over Time Was Worth it?
Description: A 5-point subject satisfaction questionnaire with the following responses: Strongly Agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree. Baseline was defined as the observation that was closest to but prior to study treatment at the baseline visit/first treatment in Study 43USSA1705. (NCT03780244). Therefore, Weeks 72 and 96 in timeframe represents timepoints of current extension study and calculated from baseline of 43USSA1705 (NCT03780244).
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Strongly Agree | 18
  Week 72: Agree | 14
  Week 72: Neither agree or disagree | 2
  Week 72: Disagree | 1
  Week 72: Strong Disagree | 0
  Week 96: Strongly Agree | 20
  Week 96: Agree | 11
  Week 96: Neither agree or disagree | 2
  Week 96: Disagree | 1
  Week 96: Strong Disagree | 1

8. Secondary Outcome: Subject Satisfaction With Treatment: Would You Say the Treatment Results Are Natural Looking?
Description: A 5-point participant satisfaction questionnaire with the following responses: Strongly Agree, Agree, Neither Agree Nor Disagree, Disagree, Strongly Disagree. Baseline was defined as the observation that was closest to but prior to study treatment at the baseline visit/first treatment in study 43USSA1705 (NCT03780244). Therefore, Weeks 72 and 96 in timeframe represents timepoints of current extension study and calculated from baseline of 43USSA1705 (NCT03780244).
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Strongly Agree | 26
  Week 72: Agree | 7
  Week 72: Neither Agree or Disagree | 1
  Week 72: Disagree | 0
  Week 72: Strongly Disagree | 1
  Week 96: Strongly Agree | 20
  Week 96: Agree | 13
  Week 96: Neither Agree or Disagree | 1
  Week 96: Disagree | 0
  Week 96: Strongly Disagree | 1

9. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Improve Your Facial Symmetry/Balance?
Description: A 5-point subject satisfaction questionnaire with the following responses: Very Satisfied, Satisfied, Neutral, Dissatisfied, Very Dissatisfied. Baseline was defined as the observation that was closest to but prior to study treatment at the baseline visit/first treatment in Study 43USSA1705 (NCT03780244). Therefore, Weeks 72 and 96 in timeframe represents timepoints of current extension study and calculated from baseline of 43USSA1705 (NCT03780244).
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Very Satisfied | 14
  Week 72: Satisfied | 14
  Week 72: Neutral (neither satisfied or dissatisfied) | 4
  Week 72: Dissatisfied | 2
  Week 72: Very Dissatisfied | 1
  Week 96: Very Satisfied | 13
  Week 96: Satisfied | 13
  Week 96: Neutral (neither satisfied or dissatisfied) | 6
  Week 96: Dissatisfied | 2
  Week 96: Very Dissatisfied | 1

10. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Make You Look the Way You Feel?
Description: as for outcome 9
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Very Satisfied | 11
  Week 72: Satisfied | 16
  Week 72: Neutral (neither satisfied or dissatisfied) | 5
  Week 72: Dissatisfied | 3
  Week 72: Very Dissatisfied | 0
  Week 96: Very Satisfied | 10
  Week 96: Satisfied | 15
  Week 96: Neutral (neither satisfied or dissatisfied) | 5
  Week 96: Dissatisfied | 4
  Week 96: Very Dissatisfied | 1

11. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Make You Look/Feel More Confident in Your Life?
Description: as for outcome 9
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Very Satisfied | 12
  Week 72: Satisfied | 16
  Week 72: Neutral (neither satisfied or dissatisfied) | 4
  Week 72: Dissatisfied | 3
  Week 72: Very Dissatisfied | 0
  Week 96: Very Satisfied | 11
  Week 96: Satisfied | 14
  Week 96: Neutral (neither satisfied or dissatisfied) | 7
  Week 96: Dissatisfied | 2
  Week 96: Very Dissatisfied | 1

12. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Improve Your Self-confidence?
Description: as for outcome 9
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Very Satisfied | 14
  Week 72: Satisfied | 13
  Week 72: Neutral (neither satisfied or dissatisfied) | 5
  Week 72: Dissatisfied | 3
  Week 72: Very Dissatisfied | 0
  Week 96: Very Satisfied | 12
  Week 96: Satisfied | 13
  Week 96: Neutral (neither satisfied or dissatisfied) | 7
  Week 96: Dissatisfied | 2
  Week 96: Very Dissatisfied | 1

13. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Improve Overall Satisfaction With Your Appearance?
Description: as for outcome 9
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Very Satisfied | 12
  Week 72: Satisfied | 17
  Week 72: Neutral (neither satisfied or dissatisfied) | 3
  Week 72: Dissatisfied | 3
  Week 72: Very Dissatisfied | 0
  Week 96: Very Satisfied | 12
  Week 96: Satisfied | 15
  Week 96: Neutral (neither satisfied or dissatisfied) | 5
  Week 96: Dissatisfied | 2
  Week 96: Very Dissatisfied | 1

14. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Make You Feel Better About Yourself?
Description: as for outcome 9
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Very Satisfied | 17
  Week 72: Satisfied | 13
  Week 72: Neutral (neither satisfied or dissatisfied) | 2
  Week 72: Dissatisfied | 3
  Week 72: Very Dissatisfied | 0
  Week 96: Very Satisfied | 13
  Week 96: Satisfied | 15
  Week 96: Neutral (neither satisfied or dissatisfied) | 4
  Week 96: Dissatisfied | 2
  Week 96: Very Dissatisfied | 1

15. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Improve Your Attractiveness?
Description: as for outcome 9
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Very Satisfied | 11
  Week 72: Satisfied | 18
  Week 72: Neutral (not satisfied or dissatisfied) | 3
  Week 72: Dissatisfied | 3
  Week 72: Very Dissatisfied | 0
  Week 96: Very Satisfied | 12
  Week 96: Satisfied | 14
  Week 96: Neutral (not satisfied or dissatisfied) | 6
  Week 96: Dissatisfied | 2
  Week 96: Very Dissatisfied | 1

16. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Make You Look Younger?
Description: as for outcome 9
Time Frame: At Weeks 72 and 96 (assessed in the current extension study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 35
Participants
  Week 72: Very Satisfied | 13
  Week 72: Satisfied | 18
  Week 72: Neutral (not satisfied or dissatisfied) | 1
  Week 72: Dissatisfied | 3
  Week 72: Very Dissatisfied | 0
  Week 96: Very Satisfied | 13
  Week 96: Satisfied | 14
  Week 96: Neutral (not satisfied or dissatisfied) | 4
  Week 96: Dissatisfied | 3
  Week 96: Very Dissatisfied | 1

17. Secondary Outcome: Number of Participants With At Least One Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence, unintended disease or injury, or untoward clinical signs of a clinical investigation in participants, whether or not related to the investigational device which included events related to the investigational product (IP) or the reference product, events related to the procedures involved and events that were anticipated as well as unanticipated. SAE: an AE resulting in death; initial or prolonged inpatient hospitalization; life-threatening experience; persistent or significant disability/incapacity; congenital anomaly. TEAE: any AEs occurring or worsening at or after first dose of IP or ongoing at time of enrollment. Baseline was defined as the observation that was closest to but prior to study treatment at the baseline visit/first treatment in Study 43USSA1705 (NCT03780244).
Time Frame: From Baseline of study 43USSA1705 (NCT03780244) up to Week 96 (assessed in the current extension study)
Population: Extension population included all participants who entered the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sculptra Aesthetic
Number analyzed (Participants) | 38
Participants
  Number of Participants with TEAEs | 24
  Number of participants with Serious TEAEs | 1

ADVERSE EVENTS:
Time Frame: From Baseline of study 43USSA1705 (NCT03780244) up to Week 96 (assessed in the current extension study)
Description: The data of this section was collected from baseline of study 43USSA1705 (NCT03780244) up to Week 96 of extension current study. Baseline was defined as the observation that was closest to but prior to study treatment at the baseline visit/first treatment in Study 43USSA1705. (NCT03780244).
Arm/Group | Sculptra Aesthetic
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 1/38
Other Adverse Events (participants affected / at risk) | 17/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sculptra Aesthetic (N=38)
Anxiety (Psychiatric disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sculptra Aesthetic (N=38)
Corona virus infection (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Headache (Nervous system disorders) | 4 (5)
Acne (Skin and subcutaneous tissue disorders) | 2 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
per site CTA

DOCUMENTS (2):
  • Study Protocol (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT04225273/Prot_003.pdf
  • Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT04225273/SAP_002.pdf